CLINICAL TRIAL: NCT06441227
Title: Phase I Clinical Study on the Safety, Tolerability and Pharmacokinetics, Pharmacodynamics and Food Effects of Single and Multiple Oral HRS-5346 Tablets in Healthy Subjects
Brief Title: Safety and Tolerance of Increased Doses of HRS-5346 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS-5346-101
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Lipoprotein Disorder Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): HRS-5346 tablets or placebo single dose
  Interventions: Drug: HRS-5346 tablets; Drug: placebo
- Part 2 (Experimental): HRS-5346 tablets or placebo single dose with food effects
  Interventions: Drug: HRS-5346 tablets; Drug: placebo
- Part 3 (Experimental): HRS-5346 tablets or placebo multiple doses
  Interventions: Drug: HRS-5346 tablets; Drug: placebo

INTERVENTIONS:
Drug: HRS-5346 tablets — Part 1: single dose. Part 2: single dose with food effects. Part 3: single dose multiple doses.
Drug: placebo — Part 1: single dose. Part 2: single dose with food effects. Part 3: single dose multiple doses.

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase I clinical study. The primary objective is to evaluate the safety, tolerability, PK, and PD of single- and multiple-dose HRS-5346 in healthy subjects, and to evaluate the food effects on PK of HRS-5346.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the specific process of the test, voluntarily participate in this test, and sign the informed consent in writing.
2. Age ≥ 18 and ≤ 55 years old on the day of signing the informed consent (including boundary value).
3. Male subjects weigh ≥ 50 kg, female subjects weigh ≥ 45kg, and BMI is in the range of 19~30 kg/m2 (including boundary values).
4. Subjects (including partners) are willing to voluntarily take effective contraceptive measures within 6 months from the time of signing the informed consent form to the last time the drug is given; the female subject's blood pregnancy test must be negative and non-lactation.
5. Normal or abnormality such as vital signs, physical examination and laboratory examination have no clinical significance.

Exclusion Criteria:

1. Those who suffer from any serious clinical diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry and metabolic abnormalities, or any other disease or medical history that can interfere with the test results or any significant laboratory abnormality that is judged by researchers to be of clinical significance.
2. Previous history of malignant tumors.
3. Those who have taken any prescription drugs, over-the-counter drugs and Chinese herbs within 14 days before taking the study drug, or within 5 half-life of the drug at the time of screening; those who plan to take non-study drugs during the trial period.
4. Those who have participated in the clinical trial of any drug or medical device within 3 months before screening, or have not been within 5 half-life of the drug before screening (when both standards are met, the standard shall be based on the long-term standard).
5. Subjects received siRNA in the past 12 months, or antisense oligonucleotide drugs in the past six months.
6. The abnormal upper limit of hypersensitive C-reactive protein during the screening period is >1.5 times the normal upper limit, or the normal upper limit of prothrombin time/international standard ratio (PT/INR), activated partial thrombin time (aPTT) > 1.25 times normal upper limit.
7. Screening for infectious diseases during the screening period (including hepatitis B virus surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, syphilis spirochete antibody).
8. 12-lead electrocardiogram abnormal and clinical significance, or electrocardiogram QT interval (QTcF) male > 450 ms, female > 470 ms.
9. The total amount of blood donated or blood loss ≥ 200 mL within 1 month before administration, or the total amount of blood donation or blood loss ≥ 400 mL within 3 months before administration, or received blood transfusion within 8 weeks.
10. Those who have a serious infection, serious trauma or major surgery within 3 months before administration; those who plan to undergo surgery within two weeks during and after the end of the trial.
11. Suspected people with a history of allergy to research drugs or any ingredients in research drugs, allergies or previous history of serious drug allergies.
12. People who have had blood collection difficulties or cannot tolerate venous punctures in the past, such as needle fainting and blood fainting.
13. Glomerular filtration rate (eGFR) is lower than GFR 60 mL/min/1.73 m2.
14. Smoke an average of ≥ 5 cigarettes per day in the first three months of administration; the average daily intake of alcohol in the first month before administration exceeded 15 grams.
15. Screening and visiting drug screening test is positive or alcohol breath test is positive.
16. Other circumstances in which the researcher believes that the subject is not suitable to participate in this experiment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Assess the incidence and severity of adverse events in healthy subjects after single and multiple doses of HRS-5346 tablets | About three months from the first medication to the evaluation

SECONDARY OUTCOMES:
Evaluation of AUC0-t of HRS-5346 in plasma and urine | About three months after the first dose
Evaluation of AUC0-inf of HRS-5346 in plasma | About three months after the first dose
Evaluation of Tmax of HRS-5346 in plasma | About three months after the first dose
Evaluation of Cmax of HRS-5346 in plasma | About three months after the first dose
Evaluation of t1/2 of HRS-5346 in plasma | About three months after the first dose
Evaluation of CL/F of HRS-5346 in plasma | About three months after the first dose
Evaluation of Vz/F of HRS-5346 in plasma | About three months after the first dose
Evaluation of Ae of HRS-5346 in urine | About three months after the first dose
Evaluation of fe of HRS-5346 in urine | About three months after the first dose
Evaluation of CLR of HRS-5346 in urine | About three months after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided